CLINICAL TRIAL: NCT02413177
Title: Augmenting Mindfulness Training Through Experience-driven Neurofeedback
Acronym: ATTEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Judson Brewer, Associate Professor, Medicine and Psychiatry, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT007922; 7R01AT007922 (NIH)
Record Dates: First submitted 2015-03-09; First posted 2015-04-09 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EEG-RTNF (Active Comparator): Group 1 will receive EEG-RTNF training from the PCC. They will attend an 8 week MBSR class. This feedback will occur at weeks 3, 4, 6 and 7.
  Interventions: Behavioral: EEG-RTNF
- EEG-no RTNF (Active Comparator): Group 2 will receive EEG (no RTNF feedback). They will attend an 8 week MBSR class. This feedback will occur at weeks 3, 4, 6 and 7.
  Interventions: Behavioral: EEG-no RTNF

INTERVENTIONS:
Behavioral: EEG-no RTNF — All EEG sessions are done on an individual basis. Group 2 will receive EEG (no RTNF) at weeks 3, 4, 6, and 7 of MBSR. At these time points, subjects will take part in a 1-hour EEG-RTNF session., comprised of six 3.5-minute runs. Each run will begin with a 30-second active baseline task in which subjects view adjectives and think about and decide if the word describes them. Following baseline, subjects will meditate for 3 to 7 minutes with EEG-RTNF. All subjects will be instructed to practice meditation during EEG-RTNF training, and to keep their eyes closed.
  Arms: EEG-no RTNF
Behavioral: EEG-RTNF — All EEG sessions are done on an individual basis. Group 1 will receive EEG-RTNF training from the PCC at weeks 3, 4, 6, and 7 of MBSR. At these time points, subjects will take part in a 1-hour EEG-RTNF session., comprised of six 3.5-minute runs. Each run will begin with a 30-second active baseline task in which subjects view adjectives and think about and decide if the word describes them. Following baseline, subjects will meditate for 3 to 7 minutes with EEG-RTNF. All subjects will be instructed to practice meditation during EEG-RTNF training, and to keep their eyes closed.
  Arms: EEG-RTNF

SUMMARY:
The overall goal of the proposed study is to develop and test real time neurofeedback (EEG-RTNF) as a tool to augment Mindfulness Based Stress Reduction (MBSR). This study is based on the theoretical model that (1) mind-wandering and self-referential processing are associated with stress, (2) meditation redirects the wandering mind toward present-centered awareness, (3) meditation also decreases activity in hubs of the default mode network (DMN) involved in mind-wandering and self-referential processing, and thus (4) meditation leading to decreased activity in these hubs should lead to reduced stress and improved health and well-being. Milestones include: (1) test whether EEG-RTNF from the PCC during meditation augments MBSR in novices; and (2) test whether MBSR with EEG-RTNF from the PCC leads to real-world outcomes in reduced stress and improved attention.

DETAILED DESCRIPTION:
Mindfulness Based Stress Reduction (MBSR) is an effective intervention for promoting positive cognitive and behavioral changes for improved health. However, MBSR delivery may be suboptimal. Recent work on potential neural mechanisms underlying the meditation practices that are core to MBSR may be utilized to improve MBSR delivery and efficacy. The investigators have shown recently that the posterior cingulate cortex (PCC), a brain region implicated in anxiety, addiction, Alzheimer's, ADHD, and other medical maladies, is selectively deactivated during three meditation practices that are core to MBSR suggesting a central role for the PCC in the neurobiology of MBSR. The investigators have also recently confirmed that PCC deactivation corresponds with the subjective experience of meditation in meditators. The proposed study will use EEG-RTNF from the PCC during meditation as an innovative strategy to augment MBSR and improve outcomes.

The task of mindfulness-the principle component of MBSR-is to maintain attention on and acceptance toward present-moment experience, and to redirect attention to one's immediate experience when it has strayed. This present-centered awareness may be considered a counterpoint to self-referential processing and mind-wandering. Consistent with a role for the PCC in mind-wandering, the PCC is specifically deactivated during three meditation practices (mindfulness of the breath, loving-kindness, and choiceless awareness) in experienced meditators compared to novices). Supporting these findings, a research study. showed that PCC deactivation during meditation correlated with a behavioral measure of attention (the Rapid Visual Information Processing Task, RVIP) in experienced meditators, suggesting that PCC deactivation is associated with improved attention in meditators. Another research study showed that the PCC is deactivated when experienced meditators mindfully view emotional images suggesting that PCC deactivation is associated with emotional stability and enhanced present-moment awareness.

EEG-RTNF is an emerging technology similar to classic biofeedback in which individuals receive moment-to-moment feedback of their brain activity during a particular task, typically by a dynamic visual display (e.g., a graph).

ELIGIBILITY:
Inclusion Criteria:

* English speakers (due to instructions provided in English)
* No history of neurological disorder
* Ability to understand the study procedures and willingness to commit to the demands of the study protocol.
* Remaining in the area for the duration of the study
* Willing to be randomized

Exclusion Criteria:

* Prior participation in an MBSR course.
* Regular meditation practice (or any other form of meditative practice, such as yoga, Tai Chi or contemplative prayer) for more than an average of 20 minutes a week within the past 2 years
* Participants with a serious psychiatric, cognitive or medical disorder which could interfere with completion of the study
* Unstable dose of psychotropic medication. Participants must be on a stable dose for the past three months
* Use of antipsychotic medication or stimulants
* Current alcohol use (>14/week or >4 drinks at any one time for a male, or >7 drinks/week or >3 drinks at any one time for a female)
* Substance abuse (high frequency and problems caused) or dependence in the past 6 months;
* Claustrophobia
* MRI incompatible implants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2015-04; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
percent signal change in the PCC as assessed by fMRI | 12 weeks
  will demonstrate that EEG-RTNF from the PCC augments MBSR as assessed by PCC deactivation during meditation

SECONDARY OUTCOMES:
Perceived stress scale (PSS) questionnaire scores, | 5 and a half month
  Show that MBSR with EEG-RTNF from the PCC leads to reduced stress and improved attention
Rapid Visual Information Processing (RVIP): %hits, | 5 and a half month
Rapid Visual Information Processing (RVIP): number of false alarms | 5 and a half month
Rapid Visual Information Processing (RVIP): % of misses | 5 and a half month
Rapid Visual Information Processing (RVIP): reaction time in milliseconds to hits | 5 and a half month
Patient Recorded Outcomes Measurement Information System (PROMIS)- 29 question scores | 5 and a half month

CONTACTS AND LOCATIONS:
Overall Officials: Judson Brewer, MD, PhD, Principal Investigator — UMass Medical School
Locations (1):
- University of Massachusetts, Worcester, Worcester, Massachusetts, United States